CLINICAL TRIAL: NCT06793579
Title: Thyroid Cancer Superior Mediastinal Lymph Node Dissection Via Lateral Cervical Approach: Exploration and Practice of a Novel Surgical Pathway
Brief Title: Lateral Approach for Mediastinal Lymph Node Dissection in Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Chongqing General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YAN-1
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer; Mediastinal Diseases; Lymph Node Metastasis
MeSH Terms: conditions — Thyroid Neoplasms; Mediastinal Diseases; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the numerous surgical approaches available for superior mediastinal lymph node dissection in thyroid cancer, many of these methods still have significant limitations. In this study, we report for the first time a novel surgical technique for superior mediastinal lymph node dissection: a thyroid cancer surgery based on a lateral cervical approach. This technique offers a new surgical option for the dissection of superior mediastinal lymph nodes in thyroid cancer.

DETAILED DESCRIPTION:
The incidence of thyroid cancer has been steadily rising over the past several decades, making it a significant focus of clinical and scientific research. Superior mediastinal lymph node metastasis, as a regional manifestation of thyroid cancer metastasis, is a clinically relevant yet underexplored phenomenon. According to previous studies, the incidence of superior mediastinal lymph node metastasis in papillary thyroid carcinoma (PTC) is approximately 6% to 12%, while in medullary thyroid carcinoma (MTC), this rate is notably higher, reaching up to 18%. Although rarer, follicular thyroid carcinoma (FTC) and anaplastic thyroid carcinoma (ATC) can also involve superior mediastinal lymph node metastasis. Despite the clinical significance of this type of metastasis, international research on its surgical management remains limited, and there is currently no standardized treatment protocol for superior mediastinal lymph node dissection in thyroid cancer patients.

At present, there are four commonly utilized surgical approaches for superior mediastinal lymph node dissection in thyroid cancer: open surgery via a cervical incision, endoscopic surgery through a cervical approach, thoracoscopic surgery, and open thoracotomy. Among these, the open surgery performed through a cervical incision is often regarded as an extension of central compartment lymph node dissection. Following the dissection of the central lymph nodes, the procedure continues downward along the trachea to remove lymph nodes situated above the right brachiocephalic artery and the left brachiocephalic vein. This approach is favored for its relatively simple learning curve, lower surgical trauma, and shorter operative time, making it a preferred method when anatomical and technical conditions allow.

However, anatomical limitations pose significant challenges to this technique. The right brachiocephalic vein lies beneath the right brachiocephalic artery, while the aortic arch are located below the left brachiocephalic vein. Even with the assistance of surgical retractors, these anatomical features often obstruct the lower portions of the lymph nodes in the superior mediastinal regions 2R and 2L, limiting surgical visibility and access. This constraint can result in incomplete lymph node dissection and, in many cases, necessitates a switch to alternative approaches such as endoscopic surgery or open thoracotomy during the procedure. Furthermore, in hospitals with limited technical expertise or surgical resources, these challenges may lead to the inability to perform superior mediastinal lymph node dissection altogether.

To address these limitations, this study seeks to propose and evaluate a novel surgical approach aimed at expanding the dissection range achievable through a cervical incision. This new technique aims to improve surgical accessibility, reduce procedural complexity, and provide a more feasible and effective option for superior mediastinal lymph node dissection in thyroid cancer. By enhancing the scope and precision of the procedure, this study aspires to contribute to the development of more standardized and widely applicable surgical strategies for the management of thyroid cancer metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who underwent thyroid cancer superior mediastinal lymph node dissection via the lateral cervical approach in our department.
2. Complete hospitalization records, ensuring that the patient's surgical records, pathological examinations, and other information are fully traceable.
3. Complete postoperative follow-up data, including complications during the follow-up period.
4. No other severe comorbidities, to avoid surgical outcome bias caused by other diseases.
5. No distant metastasis found preoperatively, or distant metastasis is still assessable for effective treatment.

Exclusion Criteria:

1. Cases with incomplete data, such as missing hospitalization records or incomplete follow-up data.
2. Systemic diseases with severe heart, lung, liver, kidney, or brain dysfunction that may affect the accuracy of data.
3. Patients with severe coagulopathy.
4. Tumor pathology indicating undifferentiated thyroid cancer, malignant lymphoma, or non-thyroid-origin tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects of this retrospective study were all patients in our department who underwent treatment with this surgical approach during the inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Number of upper mediastinal lymph nodes dissected | 1day
  Postoperative pathological records
Duration of surgery | 1day
  Described in the surgical record
Postoperative complications | 1 month
  According to the follow-up data
Surgical blood loss | 1day
  Described in the surgical record
Postoperative hospital stay | 1week
  Recorded in medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing General Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No